CLINICAL TRIAL: NCT02690142
Title: A Phase I, Partially-randomised, Partially Double-blinded, Safety, Tolerability and Pharmacokinetic Study of ABY-035 in Healthy Subjects and Psoriasis Patients
Brief Title: A Study to Investigate the Safety, Tolerability and Pharmacokinetics of ABY-035
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Affibody (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABY-035-001; 2015-004531-13 (EudraCT Number)
Record Dates: First submitted 2016-01-22; First posted 2016-02-24 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Psoriasis; Healthy Subjects
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- ABY-035 i.v. (Experimental): Part A: SAD (single ascending dose) including five different dose cohorts. ABY-035 given as intravenous injections. 6 ABY-035 and 2 placebo in each cohort.
  Interventions: Drug: Placebo; Drug: ABY-035 i.v.
- ABY-035 s.c. (Experimental): Part B: Bioavailability study where 6 subjects will receive ABY-035 as a single subcutaneous injection.
  Interventions: Drug: ABY-035 s.c.
- ABY-035 i.v. in psoriasis patients (Experimental): Part C: Up to 12 psoriasis patients will receive ABY-035 as a single intravenous injection.
  Interventions: Drug: ABY-035 i.v.
- ABY-035 s.c. in psoriasis patients (Experimental): Part D: Up to 18 patients will receive 3 or 7 biweekly doses of ABY-035 as s.c. injections
  Interventions: Drug: ABY-035 s.c.

INTERVENTIONS:
Drug: Placebo — Single dose i.v.
  Arms: ABY-035 i.v.
Drug: ABY-035 i.v. — Single dose i.v.
  Arms: ABY-035 i.v.; ABY-035 i.v. in psoriasis patients
Drug: ABY-035 s.c. — Single dose s.c.
  Arms: ABY-035 s.c.; ABY-035 s.c. in psoriasis patients

SUMMARY:
The purpose of this first-in-human study is to investigate the safety and tolerability of ABY-035 when administered intravenously and subcutaneously, to healthy volunteers and to psoriasis patients.

DETAILED DESCRIPTION:
This first in human study with ABY-035 (a novel IL-17A inhibitor (interleukin 17A)) consists of four Parts. Part A consists of a single ascending intravenous dose study with 40 healthy volunteers divided into five dose cohorts. Each group consists of 8 subjects where 6 subjects will receive ABY-035 and 2 will receive placebo. The subjects will be followed for pharmacokinetic and safety assessments up to Day 95 after dosing.

Part B of the study consists of 6 healthy volunteers who will be given a single subcutaneous dose of ABY-035. The subjects will follow the same study visit schedule as Part A.

Part C of the study will include up to 12 moderate-to-severe psoriasis patients who each patient will be given a single intravenous dose of ABY-035. The patients will follow the same study visit schedule as Part A and B.

Part D of the study will include up to 18 psoriasis patients (mild, moderate or severe). Each patient will participate in 3 or 7 biweekly dosing occasions of subcutaneously administered ABY-035. Patients will be followed regularly for safety, efficacy and pharmacokinetics for 8 weeks post-final dose.

ELIGIBILITY:
Inclusion Criteria:

Part A, Part B

* Males or females between 18 and 65 years of age
* Body mass index (BMI) between 18.0 kg/m2 and 32.0 kg/m2, inclusive. maximum body weight of 120 kg
* In good health, as determined by medical history, physical examination, vital signs assessment, 12 lead electrocardiogram (ECG) and clinical laboratory evaluations.
* Subjects will have given their written informed consent to participate in the study

In addition for Part C and D

* Males or females between 18 and 65 years of age
* Body mass index (BMI) between 18.0 kg/m2 and 39.9 kg/m2, inclusive. Minimum body weight of 45 kg
* Part C: Patients must have had a diagnosis of moderate to severe plaque type psoriasis at least 6 months prior to administration of the study drug without a documented flare within 30 days prior to Screening. Patients with concurrent psoriatic arthritis may be enrolled.
* Part D: Patients must have had a diagnosis of plaque type psoriasis (mild, moderate or severe) at least 6 months prior to administration of the study drug without a documented flare within 30 days prior to Screening. Patients with concurrent psoriatic arthritis may be enrolled.
* Part C: Have plaque type psoriasis covering at least 10% of total body surface area (BSA) at Screening and at Baseline (Day 1) and have a PASI score of 12 or greater at Screening and at Baseline (Day 1).
* Part D: Have at least one psoriatic lesion

Exclusion criteria:

Part A, Part B, Part C and Part D

* Subjects who have any clinically significant medical history, as determined by the investigator
* Subjects who smoke more than 15 cigarettes, or equivalent, per day
* Alcohol and/or drug abuse
* Positive for HIV, Hepatitis B, Hepatitis C, or tuberculosis
* Subjects who have received a live vaccination within the 3 months prior to Screening
* Subjects who are pregnant or lactating
* Subjects who do not agree to use appropriate contraception
* Subjects who have a history of anaphylaxis, drug allergy or clinically significant allergic condition (excluding non active hayfever)
* Participation in another clinical trial
* Subjects who, in the opinion of the investigator, should not participate in this study

In addition for Part C and D

* Patients who currently have non plaque forms of psoriasis (eg, erythrodermic, guttate, or pustular)
* Patients who have current drug induced psoriasis
* Have any history of any use of or have participated in clinical trials for any therapeutic agent directly targeted to any IL 17 cytokine or receptor
* Have received phototherapy within 4 weeks prior to Day 1
* Patients who have received systemic medications or treatments that could affect psoriasis or PASI evaluation (including, but not limited to, oral or injectable corticosteroids, retinoids, 1,25 dihydroxy vitamin D3 and analogues, fumaric acid esters, psoralens, anti TNF (tumour necrosis factor) biologics, anti IL 12/23 biologics, or herbal treatments), within 5 half lives prior to Day 1 (4 weeks for oral anti psoriatics, 12 weeks for psoralens and PUVA (oral psoralen with ultraviolet A), and 24 weeks for biologics)
* Patients who have used topical medications and treatments that could affect psoriasis or PASI evaluation (eg, corticosteroids, coal tar, anthralin, calcipotriene, topical vitamin D derivatives, retinoids, tazarotene, methoxsalen, and trimethyl psoralens) within 2 weeks of administration of IMP (Investigational Medicinal Product)
* Patients who have used any systemic immunosuppressants (eg, methotrexate, azathioprine, cyclosporine, 6 thioguanine, mercaptopurine, mycophenolate mofetil, hydroxyurea, or tacrolimus) within 8 weeks of administration of IMP (or 5 half lives, whichever is longer).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-02; Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values or other Adverse Events | Follow-up visit (Day 141)
  Safety is monitored by Vital signs, 12-lead ECGs, urinalysis, hematology, clinical chemistry, coagulation, proinflammatory cytokines and CRP

SECONDARY OUTCOMES:
AUC (Area Under the Concentration-time curve) of ABY-035 in healthy subjects and in patients with moderate-to-severe psoriasis through analysis of serum samples | Day 1, Day 2, Day 3, Day 4, Day 8, Day 15, Day 22, Day 29, Day 30, Day 31, Day 32, Day 43, Day 57, Day 71, Day 85, Day 95, Day 113, Day 141
t1/2 (half-life) of ABY-035 in healthy subjects and in patients with moderate-to-severe psoriasis through analysis of serum samples | Day 1, Day 2, Day 3, Day 4, Day 8, Day 15, Day 22, Day 29, Day 30, Day 31, Day 32, Day 43, Day 57, Day 71, Day 85, Day 95, Day 113, Day 141
Maximum serum concentration (Cmax) of ABY-035 in healthy subjects and in patients with moderate-to-severe psoriasis through analysis of serum samples | Day 1, Day 2, Day 3, Day 4, Day 8, Day 15, Day 22, Day 29, Day 30, Day 31, Day 32, Day 43, Day 57, Day 71, Day 85, Day 95, Day 113, Day 141
Time of maximum observed plasma concentration of ABY-035 in healthy subjects and in patients with moderate-to-severe psoriasis through analysis of serum samples | Day 1, Day 2, Day 3, Day 4, Day 8, Day 15, Day 22, Day 29, Day 30, Day 31, Day 32, Day 43, Day 57, Day 71, Day 85, Day 95, Day 113, Day 141
Time of last quantifiable plasma concentration of ABY-035 in healthy subjects and in patients with moderate-to-severe psoriasis through analysis of serum samples | Day 1, Day 2, Day 3, Day 4, Day 8, Day 15, Day 22, Day 29, Day 30, Day 31, Day 32, Day 43, Day 57, Day 71, Day 85, Day 95, Day 113, Day 141
Mean Residence Time (MRT) of ABY-035 in healthy subjects and in patients with moderate-to-severe psoriasis through analysis of serum samples | Day 1, Day 2, Day 3, Day 4, Day 8, Day 15, Day 22, Day 29, Day 30, Day 31, Day 32, Day 43, Day 57, Day 71, Day 85, Day 95, Day 113, Day 141
Total plasma clearance of ABY-035 in healthy subjects and in patients with moderate-to-severe psoriasis through analysis of serum samples | Day 1, Day 2, Day 3, Day 4, Day 8, Day 15, Day 22, Day 29, Day 30, Day 31, Day 32, Day 43, Day 57, Day 71, Day 85, Day 95, Day 113, Day 141
Absolute bioavailability (F) of ABY-035 following a single subcutaneous administration in healthy subjects. | Day 1, Day 2, Day 3, Day 4, Day 8, Day 15, Day 22, Day 29, Day 43, Day 71, Day 95
  After single subcutaneous injection
Time immediately prior to first quantifiable concentration of ABY-035 following a single subcutaneous administration in healthy subjects. | Day 1, Day 2, Day 3, Day 4, Day 8, Day 15, Day 22, Day 29, Day 43, Day 71, Day 95
  After single subcutaneous injection
Volume of distribution during the terminal elimination phase of ABY-035 in healthy subjects and in patients with moderate-to-severe psoriasis through analysis of serum samples | Day 1, Day 2, Day 3, Day 4, Day 8, Day 15, Day 22, Day 29, Day 30, Day 31, Day 32, Day 43, Day 57, Day 71, Day 85, Day 95, Day 113, Day 141
Volume of distribution at steady state of ABY-035 in healthy subjects and in patients with moderate-to-severe psoriasis through analysis of serum samples | Day 1, Day 2, Day 3, Day 4, Day 8, Day 15, Day 22, Day 29, Day 30, Day 31, Day 32, Day 43, Day 57, Day 71, Day 85, Day 95, Day 113, Day 141
Clinical efficacy of ABY-035, using PASI (Psoriasis Area and Disease Index) response, following single dose intravenous administration in patients with moderate-to-severe psoriasis. | Screening, Day -1, Day 2, Day 8, Day 15, Day 17, Day 22, Day 29, Day 31, Day 43, Day 71, Day 57, Day 85, Day 95, Day 113, Day 123, Day 141, Day 151
Immunogenicity of ABY-035 in healthy subjects and in patients with moderate-to-severe psoriasis | Day -1, Day 1, Day 15, Day 29, Day 57, Day 85, Day 95, Day 113, Day 141
  Measurement of the occurrence of anti-drug antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Sunu Valasseri, MBBS, MSc, Principal Investigator — Covance Ltd
Locations (4):
- United Kingdom (4):
  - Covance Clinical Research Unit Ltd., Leeds
  - Covance and Royal Liverpool University Hospital Clinical Research Unit, Liverpool
  - Imperial Centre for Translational and Experimental Medicine Imperial College Healthcare NHS Trust Hammersmith Hospital, London
  - Medicines Evaluation Unit Ltd, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klint S, Feldwisch J, Gudmundsdotter L, Dillner Bergstedt K, Gunneriusson E, Hoiden Guthenberg I, Wennborg A, Nyborg AC, Kamboj AP, Peloso PM, Bejker D, Frejd FY. Izokibep: Preclinical development and first-in-human study of a novel IL-17A neutralizing Affibody molecule in patients with plaque psoriasis. MAbs. 2023 Jan-Dec;15(1):2209920. doi: 10.1080/19420862.2023.2209920. PMID 37184136